CLINICAL TRIAL: NCT05008887
Title: Efficacy of Fractional CO2 Laser-assisted Cutaneous Delivery of Methotrexate Versus 5-fluorouracil in Stable Non-segmental Vitiligo
Brief Title: Fractional CO2 Laser-assisted Cutaneous Delivery of Methotrexate Versus 5-fluorouracil in Stable Non-segmental Vitiligo
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Mohamed, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTXVITILIGO
Record Dates: First submitted 2021-08-10; First posted 2021-08-17 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Methotrexate; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fractional CO2 laser and topical methotrexate solution (Experimental): In all patients, the selected patches of vitiligo will be treated with fractional CO2 laser for 3 sessions at one-month intervals.
  In each patient, two patches or their duplicates (if small sized) will be subjected first to fractional CO2 laser treatment at two different energies (half the number of selected patches will be treated with 50 mJ-energy "with the aim to use laser more as a delivery system to drug solution", and the other half will be treated with 100mJ-energy "with the aim to use laser as both therapeutic and delivery system" , followed by topical application of methotrexate solution (2.5% concentration "vial 50mg/2ml" using insulin syringe as 0.1 ml at 1 cm-intervals with a maximum volume of 2 ml per session). Then gentle massage will be done and after about 10 minutes, an occlusive dressing will be applied for 24 hours after the session.
  In all patients, the selected patches of vitiligo will be treated with fractional CO2 laser for 3 sessions at one-month intervals.
  Interventions: Drug: Methotrexate; Device: Fractional CO2 laser
- Fractional CO2 laser and topical 5-fluorouracil solution (Active Comparator): In all patients, the selected patches of vitiligo will be treated with fractional CO2 laser for 3 sessions at one-month intervals.
  In each patient, two patches or their duplicates (if small sized) will be subjected first to fractional CO2 laser treatment at two different energies (half the number of selected patches will be treated with 50 mJ-energy "with the aim to use laser more as a delivery system to drug solution", and the other half will be treated with 100mJ-energy "with the aim to use laser as both therapeutic and delivery system" , followed by topical application of 5-fluorouracil solution 5% concentration "vial 250mg/5ml" using insulin syringe as 0.1 ml at 1 cm-intervals with a maximum volume of 2 ml per session). Then gentle massage will be done and after about 10 minutes, an occlusive dressing will be applied for 24 hours after the session.
  In all patients, the selected patches of vitiligo will be treated with fractional CO2 laser for 3 sessions at one-month intervals.
  Interventions: Drug: 5-fluorouracil; Device: Fractional CO2 laser

INTERVENTIONS:
Drug: Methotrexate — Fractional CO2 laser-assisted cutaneous delivery of methotrexate solution in stable, non-segmental vitiligo
  Arms: Fractional CO2 laser and topical methotrexate solution
Drug: 5-fluorouracil — Fractional CO2 laser-assisted cutaneous delivery of 5-fluorouracil solution in stable, non-segmental vitiligo
  Arms: Fractional CO2 laser and topical 5-fluorouracil solution
Device: Fractional CO2 laser — Fractional CO2 laser-assisted cutaneous delivery of methotrexate and 5-fluorouracil solution in stable, non-segmental vitiligo

SUMMARY:
Vitiligo is a common acquired, depigmenting skin disease that affect the patient's psychological state and quality of life.

DETAILED DESCRIPTION:
Vitiligo is a common acquired, depigmenting skin disease that affect the patient's psychological state and quality of life.

Regarding treatment of vitiligo, several modalities are available but none are completely satisfactory. Recently, fractional carbon dioxide (CO2) laser has been introduced as an add-on treatment for vitiligo.

Fractional CO2 laser acts by stimulating the release of cytokines and growth factors that act as mitogens for melanogenesis. Also, microscopic ablative zones produced by it promote the trans-epidermal penetration of topical agents, providing additional benefits for re-pigmentation.

Recently topical methotrexate 1% gel was used in a case report of vitiligo and was applied to a single patch twice daily for 12 weeks with significant improvement in pigmentation without local or systemic side effects during the course of therapy. Thus, it may prove to be an important steroid sparing agent in treatment of vitiligo.

As methotrexate is a large, hydrophilic molecule that does not penetrate intact skin, several drug delivery systems are being developed e.g. nano-vehicle preparations and laser-assisted delivery. One study has evaluated fractional Erbium laser-assisted delivery of topical methotrexate in porcine skin and found that methotrexate distribution and concentration in the mid-dermis was facilitated by ablative fractional laser, suggesting that ablative fractional laser-assisted topical methotrexate-delivery may be an appropriate alternative to systemic methotrexate for some skin disorders.

Ablative fractional laser-assisted delivery of topical 5-fluorouracil has been used in vitiligo in several studies with good results.

Serum interleukin-23 levels were significantly higher in vitiligo patients as compared with controls.

ELIGIBILITY:
Inclusion Criteria:

The patients will be enrolled in the study if they have:

* Non-segmental vitiligo
* Stable disease (a patient reporting no new lesions, no progression of existing lesions, and absence of Koebner phenomenon during the past 1 year)

Exclusion Criteria:

1. History of skin cancers, keloid, hypertrophic scars or photosensitivity.
2. Use of any topical medications, phototherapy, or laser for vitiligo within 1 month prior to enrollment.
3. Renal, hepatic, hematological or debilitating chronic diseases.
4. Active inflammation or infection at site of treatment.
5. Pregnant and lactating females.
6. Age under 18 years old.
7. Segmental vitiligo, active or extensive disease.
8. Unrealistic expectation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation | 6 month (3 months of treatment and 3 months for follow up after last treatment)
  Photographic evaluation
  * Patients will be evaluated by digital photographs at baseline, before each session and monthly for 3 months after the last session to evaluate the therapeutic response.
  * Two non-treating blinded dermatologists will be asked to record percentage of improvement in the treated patches for each patient after completion of the treatment by comparing before and after digital photographs. The re-pigmentation response will be expressed qualitatively using a quartile grading scale (grade 0 = no improvement; 1, 1-25% = minimal; 2, 26-50% = moderate; 3, 51-75% = good; and 4, >75% = excellent).
  Quantitative assessment by the point counting technique:
  Quantitative assessment will be done by calculating the area of depigmentation in vitiliginous patches using a simple point counting method at baseline, before each session and at the final evaluation.
  The percentage reduction in lesion size will be then calculated.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lai YC, Yew YW, Kennedy C, Schwartz RA. Vitiligo and depression: a systematic review and meta-analysis of observational studies. Br J Dermatol. 2017 Sep;177(3):708-718. doi: 10.1111/bjd.15199. Epub 2017 Jul 23. PMID 27878819
- [Background] Agarwal K, Podder I, Kassir M, Vojvodic A, Schwartz RA, Wollina U, Valle Y, Lotti T, Rokni GR, Grabbe S, Goldust M. Therapeutic options in vitiligo with special emphasis on immunomodulators: A comprehensive update with review of literature. Dermatol Ther. 2020 Mar;33(2):e13215. doi: 10.1111/dth.13215. Epub 2020 Jan 12. PMID 31891450
- [Background] Kim HJ, Hong ES, Cho SH, Lee JD, Kim HS. Fractional Carbon Dioxide Laser as an "Add-on" Treatment for Vitiligo: A Meta-analysis with Systematic Review. Acta Derm Venereol. 2018 Feb 7;98(2):180-184. doi: 10.2340/00015555-2836. PMID 29110015
- [Background] Shin J, Lee JS, Hann SK, Oh SH. Combination treatment by 10 600 nm ablative fractional carbon dioxide laser and narrowband ultraviolet B in refractory nonsegmental vitiligo: a prospective, randomized half-body comparative study. Br J Dermatol. 2012 Mar;166(3):658-61. doi: 10.1111/j.1365-2133.2011.10723.x. Epub 2012 Jan 19. PMID 22050270
- [Background] Abdelmaksoud A, Dave DD, Lotti T, Vestita M. Topical methotrexate 1% gel for treatment of vitiligo: A case report and review of the literature. Dermatol Ther. 2019 Sep;32(5):e13013. doi: 10.1111/dth.13013. Epub 2019 Jul 16. PMID 31265164
- [Background] Aickara D, Bashyam AM, Pichardo RO, Feldman SR. Topical methotrexate in dermatology: a review of the literature. J Dermatolog Treat. 2022 Feb;33(1):512-517. doi: 10.1080/09546634.2020.1770170. Epub 2020 May 25. PMID 32412810
- [Background] Taudorf EH, Lerche CM, Vissing AC, Philipsen PA, Hannibal J, D'Alvise J, Hansen SH, Janfelt C, Paasch U, Anderson RR, Haedersdal M. Topically applied methotrexate is rapidly delivered into skin by fractional laser ablation. Expert Opin Drug Deliv. 2015 Jul;12(7):1059-69. doi: 10.1517/17425247.2015.1031216. Epub 2015 Apr 20. PMID 25893560
- [Background] Doghaim NN, El-Tatawy RA, Ismail MA, Ali DAM, El Attar YA. Study the effect of erbium:YAG laser plus topical 5-flurouracil in stable vitiligo resistant to NB-UVB phototherapy. J Cosmet Dermatol. 2020 Jan;19(1):122-130. doi: 10.1111/jocd.13134. Epub 2019 Oct 1. PMID 31571367
- [Background] Anbar TS, Westerhof W, Abdel-Rahman AT, Ewis AA, El-Khayyat MA. Effect of one session of ER:YAG laser ablation plus topical 5Fluorouracil on the outcome of short-term NB-UVB phototherapy in the treatment of non-segmental vitiligo: a left-right comparative study. Photodermatol Photoimmunol Photomed. 2008 Dec;24(6):322-9. doi: 10.1111/j.1600-0781.2008.00385.x. PMID 19000191
- [Background] Vaccaro M, Cannavo SP, Imbesi S, Cristani M, Barbuzza O, Tigano V, Gangemi S. Increased serum levels of interleukin-23 circulating in patients with non-segmental generalized vitiligo. Int J Dermatol. 2015 Jun;54(6):672-4. doi: 10.1111/ijd.12392. Epub 2014 Nov 27. PMID 25427848
- [Background] Kadry M, Tawfik A, Abdallah N, Badawi A, Shokeir H. Platelet-rich plasma versus combined fractional carbon dioxide laser with platelet-rich plasma in the treatment of vitiligo: a comparative study. Clin Cosmet Investig Dermatol. 2018 Nov 8;11:551-559. doi: 10.2147/CCID.S178817. eCollection 2018. PMID 30510437